CLINICAL TRIAL: NCT03555604
Title: Evaluation of the Effect of Body Mass Index on Gastric Volume With Ultrasound in Term Pregnant Women
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor Department of Anesthesiology and Perioperative Medicine, Augusta University
Other Study IDs: 1184342
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy Related; Aspiration; Airway Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scheduled cesarean section: Gastric ultrasound in term pregnant patients to correlate with NPO time in relation to body mass index
  Interventions: Diagnostic Test: Gastric ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — Gastric ultrasound to measure antrum cross sectional area

SUMMARY:
This study seeks to determine if a relationship exists between gastric antrum cross-sectional area measured using ultrasound and BMI in term pregnant women (>37 weeks gestation).

DETAILED DESCRIPTION:
After approval by the Institutional Review Board, the investigators will obtain consent from patients. The consent will be obtained by the authorized personnel as per protocol, in which the investigators will explain to the patient the procedure, benefit, risk, cost and, confidentiality. The investigators plan to get the consent immediately after the patient arrived at the unit to avoid any interference with the delivery process. If the patient needs to go to an emergency cesarean section. This patient is not going to be included in the study. A gastric ultrasound with a low frequency (1-5 Hz) curvilinear array transducer using a Philips (CX-50) (Bothell, WA. USA) with image compounding technology, will be performed in each patient. The ultrasound procedure will be performed in the supine position and in a semi-recumbent right lateral position. The antrum will be identified in the sagittal plane between the liver, pancreas and aorta between peristaltic contractions. The ultrasound will be performed in each patient, in each position by three operators: two staff anesthesiologists and an anesthesia resident in presence of a medical student who will make sure that the standards for the procedure are uniform between operators (three images will be recorded by each operator per position in each patient). A qualitative assessment will be initially made, consisting of three grades: Grade 0, no fluid evidenced; Grade 2, clear fluid is evidenced only in right lateral decubitus position, and Grade 3, fluid is evidenced in both positions. Quantitative measurement of the cross-sectional area of the antrum (CSA) will be done by means of free tracing calipers. The full-thickness of the gastric wall will be included in the measurement and the average from the three images of each operator will be recorded. CSA will be calculated using the following formula:

CSA =(π x mean anteroposterior diameter x mean longitudinal diameter)/4

In addition to qualitative and quantitative ultrasound measures, the investigators will record demographic variables including age, BMI, weeks of gestation, gravity and parity.

The investigators plan to evaluate the existence of a relationship between cross-sectional area of the antrum (CSA) and BMI in term pregnant women using measurements of the CSA taken with free tracing calipers in ultrasound

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients >37 weeks of gestation
2. Age older than 18 years
3. NPO status >6 hours

Exclusion Criteria:

1. Unwillingness to participate in the study
2. Diagnosis of upper gastrointestinal disease
3. Episode of vomiting within the last 6 hours
4. Patients taking gastric pro-kinetic medications
5. Diabetes mellitus
6. Prior gastric, esophageal or upper abdominal surgery
7. Allergy to US gel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Term pregnant patients scheduled for cesarean section
Study Population: Term pregnant patients scheduled for cesarean section, who meet inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Cross sectional area of gastric antrum | 10 minutes
  Cross sectional area of gastric antrum

SECONDARY OUTCOMES:
BMI | 10 minutes
  Body mass index
Fasting time | 8 hours
  NPO status

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No